CLINICAL TRIAL: NCT06076395
Title: The Effect of Volume Controlled Versus Pressure Ventilation on Anesthesia Induced Lung Atelectasis in Pediatrics Using Laryngeal Mask Airway (LMA )During Cardiac Catheterization. A Prospective Randomized Study.
Brief Title: Volume Versus Pressure Ventilation on Lung Atelectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Dalia Saad Abd-El Kader, assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MS-96-2023
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Congenital Defects
Keywords: pediatric cardiac catheterization; lung ultrasound score; lung atelectasis; LMA
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: For group A pressure control ventilation will be adjusted as follows:
  Inspiratory pressure will be adjusted to achieve an expired tidal volume of 7 ml/Kg, respiratory rate will be adjusted to achieve an end ETCO2 at 32-35 mmHg, inspiratory to expiratory ratio at 1:2, PEEP at 4 cm H 2 O and FiO2 at 0.5 providing that the maximum airway pressure will be limited to 25 cmH2O.
  For group B volume control ventilation will be adjusted as follows:
  tidal volume (VT) adjacent to 7 ml/Kg, respiratory rate will be adjusted to achieve an end ETCO2 at 32-35 mmHg and I/E at: 1:2 and positive end expiratory pressure (PEEP)at 4 cmH2O and FiO2 at 0.5.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomly allocated by a computer-generated list (www.randomization.com) into one of the study groups in the day of the study . The randomization sequence will be concealed in sealed envelopes and will be opened by an independent nurse. The data collector and data analysis will be blind to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A pressure control ventilation (Experimental): Inspiratory pressure was adjusted to achieve an expired tidal volume of 7 ml/Kg, respiratory rate was adjusted to achieve an end ETCO2 at 32-35 mmHg, inspiratory to expiratory ratio at 1:2, PEEP at 4 cm H2O and FiO2 at 0.5 providing that the maximum airway pressure was limited to 25 cmH2O.
  Interventions: Device: LMA (Laryngeal Mask Airway)
- Group B volume control ventilation (Experimental): VT adjacent to 7 ml/Kg, respiratory rate was adjusted to achieve an end ETCO2 at 32-35 mmHg and I/E at: 1:2 and PEEP at 4 cm H2O and FiO2 at 0.5.
  Interventions: Device: LMA (Laryngeal Mask Airway)

INTERVENTIONS:
Device: LMA (Laryngeal Mask Airway) — Pressure controlled versus Volume controlled ventilation using LMA
  Other Names: Lung Ultrasound

SUMMARY:
This prospective randomized comparative study, to assess post-operative lung atelectasis by comparing calculated lung score using ultrasound between pediatric patients intubated with LMA (laryngeal mask airway) under volume versus pressure controlled modes of ventilation.

DETAILED DESCRIPTION:
The initial US scanning will be done prior to the induction of anesthesia. Induction of anesthesia using 4% sevoflurane. Adequate size LMA will be inserted after adequate depth of anesthesia adjusted.

Group A (n=25): will receive pressure-controlled ventilation (PCV). Group B (n=25): will receive volume-controlled ventilation (VCV).

US scanning and Arterial blood gases at the following:

* T1(After maintenance of anesthesia).
* T2 (One minute after applying groin bandage and before extubation).
* T3 (10 minutes after extubation and resumption of adequate regular breathing).
* T4 (30 min post extubation).

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients undergoing cardiac catheterization procedures. Age from 2 years to 6 years of both sexes.

Exclusion Criteria:

* Lung score at different times.
* Age <2 years and >6 years.
* Preoperative mechanical ventilation.
* Heart failure (any inotropic support infusion).
* Patients with any lung diseases( acute respiratory disease, pulmonary or lung
* diseases).
* Lung consolidation score ≥ 2 before insertion of LMA.
* Any contraindication for LMA insertion (risk for aspiration, and/or airway
* obstruction below the larynx.)
* Procedures exceeding 120 mins duration.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Post operative incidence of Lung atelectasis immediate post-removal of LMA. | immediated post removal of LMA
  calculate lung score using lung ultrasound

SECONDARY OUTCOMES:
Correlation between lung score and PaO2 /FiO2 ratio | From the preoperative period (T0) to 30 minutes post-extubation
  Arterial blood gases (ABG) in different time

CONTACTS AND LOCATIONS:
Overall Officials: Amel Hanfy Abo El- Ela, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- Dalia Saad, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hedenstierna G. Airway closure, atelectasis and gas exchange during anaesthesia. Minerva Anestesiol. 2002 May;68(5):332-6. PMID 12029240
- [Background] Stefanik E, Drewnowska O, Lisowska B, Turek B. Causes, Effects and Methods of Monitoring Gas Exchange Disturbances during Equine General Anaesthesia. Animals (Basel). 2021 Jul 9;11(7):2049. doi: 10.3390/ani11072049. PMID 34359177
- [Background] Chiumello D, Mongodi S, Algieri I, Vergani GL, Orlando A, Via G, Crimella F, Cressoni M, Mojoli F. Assessment of Lung Aeration and Recruitment by CT Scan and Ultrasound in Acute Respiratory Distress Syndrome Patients. Crit Care Med. 2018 Nov;46(11):1761-1768. doi: 10.1097/CCM.0000000000003340. PMID 30048331
- [Background] Rodriguez-Fanjul J, Corsini I, Orti CS, Bobillo-Perez S, Raimondi F. Lung ultrasound to evaluate lung recruitment in neonates with respiratory distress (RELUS study). Pediatr Pulmonol. 2022 Oct;57(10):2502-2510. doi: 10.1002/ppul.26066. Epub 2022 Jul 12. PMID 35792663
- [Background] Li X, Liu B, Wang Y, Xiong W, Zhang Y, Bao D, Liang Y, Li L, Liu G, Jin X. The effects of laryngeal mask airway versus endotracheal tube on atelectasis in patients undergoing general anesthesia assessed by lung ultrasound: A protocol for a prospective, randomized controlled trial. PLoS One. 2022 Sep 9;17(9):e0273410. doi: 10.1371/journal.pone.0273410. eCollection 2022. PMID 36084154
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376